CLINICAL TRIAL: NCT02821260
Title: Clinical Evaluation of the Efficacity of Epilepsy Surgery in Infants and Children
Acronym: PEPSI
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CBU_2015_29
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The Pediatric Neurosurgery Service of the Rothschild Foundation (Paris) is the French leader center for surgery of epilepsy in infants and children.

Postoperative follow-up of these children is performed during medical and neurosurgical consultations in order to assess the frequency of attacks and to reduce medication.

On average, two postoperative consultations are carried out between 3 and 5 months and between 12 and 18 months. Beyond 18 months, some children may benefit from long-term monitoring at this center, but most children are followed by their neurologist .

Therefore, the center has no rigorous and systematic collection of standardized data on the outcome of these patients.

The purpose of this study is to evaluate the efficacy of the epilepsy surgery in children with a monitoring of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Child treated surgically for epilepsy at the Rothschild Foundation (Paris, France)

Exclusion Criteria:

* Parental opposition to the participation of their child to the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric epilepsy requiring surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of seizures | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France